CLINICAL TRIAL: NCT03333317
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Orally Administered Lumicitabine (JNJ-64041575) Regimens in Hospitalized Infants and Children Aged 28 Days to 36 Months Infected With Respiratory Syncytial Virus
Brief Title: A Study to Evaluate the Antiviral Activity, Clinical Outcomes, Safety, Tolerability, and Pharmacokinetics of Orally Administered Lumicitabine (JNJ-64041575) Regimens in Hospitalized Infants and Children Aged 28 Days to 36 Months Infected With Respiratory Syncytial Virus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108367; 2017-001862-56 (EudraCT Number); 64041575RSV2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Respiratory Syncytial Viruses
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (Low-Dose Lumicitabine) (Experimental): Participants will receive a single 40 milligram per kilogram (mg/kg) loading dose (LD) (Dose 1) followed by nine 20 mg/kg maintenance doses (MDs) (Doses 2 to 10) of lumicitabine twice daily up to Day 5/6.
  Interventions: Drug: Lumicitabine
- Regimen B (High-Dose Lumicitabine) (Experimental): Participants will receive a single 60 mg/kg LD (Dose 1) followed by nine 40 mg/kg MDs (Doses 2 to 10) of lumicitabine twice daily up to Day 5/6.
  Interventions: Drug: Lumicitabine
- Regimen C (Placebo) (Placebo Comparator): Participants will receive either a single 40 mg/kg placebo LD (Dose 1) followed by nine 20 mg/kg maintenance dose (MDs) (Doses 2 to 10) of placebo twice daily or single 60 mg/kg placebo LD (Dose 1) followed by nine 40 mg/kg placebo MDs (Doses 2 to 10), twice daily up to Day 5/6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumicitabine — Participants will receive oral administration of lumicitabine.
  Other Names: ALS-008176; JNJ-64041575
  Arms: Regimen A (Low-Dose Lumicitabine); Regimen B (High-Dose Lumicitabine)
Drug: Placebo — Participants will receive oral administration of matching placebo.
  Arms: Regimen C (Placebo)

SUMMARY:
The purpose of this study is to determine in hospitalized infants and children who are infected with respiratory syncytial virus (RSV) the dose-response relationship of multiple regimens of lumicitabine on antiviral activity based on nasal RSV shedding using quantitative real-time reverse transcriptase polymerase chain reaction (qRT-PCR).

DETAILED DESCRIPTION:
RSV is a leading cause of lower respiratory tract disease in infants. Most infants and children who get RSV recover fully after 1-2 weeks, but RSV infection can sometimes worsen and may lead to hospitalization and admission into an intensive care unit. The main purpose of this study is to learn how well the study drug (lumicitabine, also known as JNJ-64041575 or ALS-008176) works, how the human body handles the study drug, which dose of the study drug is effective for treatment of RSV infection in infants/children and how safe it is compared to a placebo (placebo looks just like lumicitabine [given in same way] but has no effect against RSV). Approximately up to 180 participants aged between 28 days to 36 months and hospitalized with RSV infection will take part in this world-wide study.

ELIGIBILITY:
Inclusion Criteria:

* Participants hospitalized (or in emergency room [ER]) at the time of randomization and unlikely to be discharged for the first 24 hours after randomization
* Participants diagnosed with respiratory syncytial virus (RSV) infection using a polymerase chain reaction (PCR)-based molecular diagnostic assay, with or without co-infection with another respiratory pathogen (respiratory virus or bacteria)
* Participants who have an acute respiratory illness with signs and symptoms consistent with a viral infection (for example, fever, cough, nasal congestion, runny nose, sore throat, myalgia, lethargy, shortness of breath, or wheezing) with onset less than or equal to <=5 days from the anticipated time of randomization. Onset of symptoms is defined as the first time (within 1 hour) the parent(s)/caregiver(s) becomes aware of respiratory or systemic symptoms of RSV infection
* With the exception of the symptoms related to the RSV infection or defined comorbid condition for severe RSV disease (prematurity at birth [participant's gestational age was less than {<}37 weeks; for infants <1 year old at randomization], bronchopulmonary dysplasia, congenital heart disease, other congenital diseases, Down syndrome, neuromuscular impairment, or cystic fibrosis), participant must be medically stable on the basis of physical examination, medical history, vital signs/peripheral capillary oxygen saturation (SpO2), and electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying condition in the study population and/or the RSV infection. This determination must be recorded in the participant's source documents and initialed by the investigator. Participants with comorbidities will be allowed to be enrolled once the Independent Data Monitoring Committee (IDMC) has reviewed the pharmacokinetic (PK) and safety data of the highest dose that will be used in this study and once the IDMC has recommended opening recruitment to this group. Sites will be notified when the restriction is lifted
* The participant's estimated glomerular filtration rate (eGFR) is not below the lower limit of normal for the participant's age

Exclusion Criteria:

* Participants who are not expected to survive for more than 48 hours
* Participants who have had major thoracic or abdominal surgery in the 6 weeks prior to randomization
* Participants who have a known or suspected immunodeficiency (except immunoglobulin A [IgA] deficiency), such as a known human immunodeficiency virus infection
* Participants being treated with extracorporeal membrane oxygenation
* Participant receiving chronic oxygen therapy at home prior to admission
* Participants who have a poorly functioning gastrointestinal tract (that is, unable to absorb drugs or nutrition via enteral route)

Ages: 28 Days to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- United States (6):
  - MemorialCare Research Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - The Children's Mercy Hospital, Kansas City, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - West Virginia University, Morgantown, West Virginia
  - American Family Children's Hospital, Madison, Wisconsin
- Huderf, Brussels, Belgium
- McMaster Children's Hospital, Hamilton, Ontario, Canada
- Hungary (3):
  - Heim Pal Gyermekkorhaz, Borgyogyaszati Osztaly, Budapest
  - Velkey László Gyermekegészségügyi Központ, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
- Japan (16):
  - National Hospital Organization Fukuoka Hospital, Fukuoka
  - Fukuoka Children's Hospital, Fukuoka
  - National Hospital Organization Fukuyama Medical Center, Fukuyama
  - Fukuyama City Hospital, Fukuyama
  - JA Hiroshima General Hospital, Hatsukaichi
  - Hirosaki National Hospital, Hirosaki
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - National Hospital Organization Kokura Medical Center, Kitakyushu
  - National Hospital Organization Niigata National Hospital, Niigata
  - Nakano Children's Hospital, Osaka
  - Takatsuki General Hospital, Osaka
  - NHO Beppu Medical Center, Ōita
  - Ota Memorial Hospital, Ōta-ku
  - NHO Saitama National Hospital, Saitama
  - Gunma Children's Medical Center, Shibukawa
  - Shikoku Medical Center for Children and Adults, Zentsujichó
- Poland (2):
  - Plejady Medical Center, Malopolska
  - Specialistic Hospital Center for Mother and Child, Poznan

REFERENCES:
- [Derived] Oey A, McClure M, Symons JA, Chanda S, Fry J, Smith PF, Luciani K, Fayon M, Chokephaibulkit K, Uppala R, Bernatoniene J, Furuno K, Stanley T, Huntjens D, Witek J; 503 and RSV2004 Study Groups. Lumicitabine, an orally administered nucleoside analog, in infants hospitalized with respiratory syncytial virus (RSV) infection: Safety, efficacy, and pharmacokinetic results. PLoS One. 2023 Jul 19;18(7):e0288271. doi: 10.1371/journal.pone.0288271. eCollection 2023. PMID 37467213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On 17 October 2018, the study was stopped prematurely by the sponsor as a precautionary measure, to allow further evaluation and assessment of the new nonclinical pharmacokinetics (PK) and safety findings and determine their relevance to human studies.
Pre-assignment Details: Total 7 participants were randomized to receive lumicitabine or placebo.
Groups:
- Placebo: Participants received a single dose of lumicitabine-40 milligrams/kilogram (mg/kg) matched placebo as a loading dose (LD) (Dose 1) followed by 9 maintenance dose (MD) of lumicitabine-20 mg/kg matched placebo twice a day or a single dose of lumicitabine-60 mg/kg matched placebo LD (Dose 1) followed by nine lumicitabine-40 mg/kg matched placebo MD (Dose 2 to 10).
- Lumicitabine 40/20 mg/kg LD/MD: Participants received a single dose of lumicitabine-40 mg/kg as LD (Dose 1) followed by 9 MD doses of lumicitabine 20 mg/kg twice a day.
- Lumicitabine 60/40 mg/kg LD/MD: Participants received a single dose of lumicitabine-60 mg/kg as LD (Dose 1) followed by 9 MD doses of lumicitabine 40 mg/kg twice a day.
Period: Overall Study
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD | Total
Number analyzed (Participants) | 3 | 1 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: months] | 16 (13.08) | 17 | 6.3 (2.52) | 12 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 3 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 1 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Respiratory Syncytial Virus (RSV) Viral Load
Description: AUC of RSV viral load was measured by quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) assay of the mid-turbinate nasal swab.
Time Frame: Day 1 to 7: Predose, 0.25 and 2 hours postdose
Population: As study was terminated early with fewer participants than planned, data for this outcome measure was not collected and analyzed.
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Emergent Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. All AEs reported during treatment or follow-up were considered emergent and were included in the analysis.
Time Frame: Up to 28 days
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 3 | 1 | 3

3. Secondary Outcome: Number of Participants With Clinically Significant Physical Examinations Abnormalities
Description: The number of participants with clinically significant physical examination (respiratory system, nose, ear, throat, facial and neck lymph nodes, and skin examination) abnormalities that emerged after treatment initiation was reported.
Time Frame: Up to 28 days
Population: Randomized or Treated set was defined as all participants who were in Randomized Analysis Set (all randomized participants with a randomization date at or before the date of the first intake of medication, or with a randomization date and a missing date for first medication intake, analyzed as randomized) and/or all participants treated (AST) set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 2 | 1 | 1

4. Secondary Outcome: Number of Participants With Emergent Clinical Relevant Vital Signs Abnormalities
Description: The number of participants with emergent clinically relevant vital signs (temperature, pulse rate, respiratory rate, diastolic blood pressure, systolic blood pressure, oxygen saturation) abnormalities that emerged after treatment initiation reported. An abnormality was considered emergent in a particular phase if it is worse than baseline. If baseline is missing, the abnormality is always considered as emergent. A shift from 'abnormally low' at baseline to 'abnormally high' post baseline (or vice versa) was also emergent.
Time Frame: Up to 28 days
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants
  Systolic Blood Pressure (Abnormally high) | 2 | 1 | 1
  Diastolic Blood Pressure (Abnormally high) | 1 | 1 | 0
  Pulse Rate (Abnormally high) | 1 | 1 | 1
  Respiratory Rate (Abnormally high) | 0 | 0 | 1
  Temperature (High) | 1 | 0 | 1
  Oxygen Saturation (Abnormally low) | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: The number of participants with ECG (QT, and QTc intervals) abnormalities reported.
Time Frame: Up to 28 days
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants
  QT Duration | 1 | 0 | 0
  QTcB: Bazett's Correction Formula | 0 | 0 | 0
  QTcF: Fridericia's Correction Formula | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Worst Emergent Laboratory Abnormalities (Division of Microbiology and Infectious Diseases [DMID] Toxicity Grades)
Description: Number of participants with Laboratory (hematology, serum chemistry, and urinalysis) abnormalities reported based on DMID toxicity grading scale. DMID toxicity grades ranges from 1 to 4. Grade 0 is normal and not meeting the criteria of Grade 1-4. Hb: Grade 1: for 22-35 days old- 9.5-10.5 gram per deciliter (g/dL); for 36-60 days old- 8.5-9.4 g/dL; for 61-90 days old- 9.0-9.9 g/dL; Hb: Grade 2: for 22-35 days old- 8.0-9.4 g/dL, for 36-60 days old- 7.0-8.4 g/dL; for 61-90 days old- 7.0-8.9 g/dL. ALT: Grade 1- 1.1 - <2.0*Upper limit of normal (ULN); Creatinine: Grade 2- 1.8-2.4 milligram per deciliter (mg/dL); Hyperkalemia: Grade 1- 3.0-3-5 milliequivalents per Liter (mEq/L); ANC: Grade 1: for 7-60 days old- 1200-1800/ millimeter cube(mm^3); for 61-90 days old- 750-1200/mm^3; ANC: Grade 3: for 7-60 days old- 500-899/mm^3, for 61-90 days old- 250-399/mm^3; ANC: Grade 4- for 7-60 days old <500/mm^3, for 61-90 days old- <250/mm^3; Platelets: Grade 3: 25000 - 49999/mm^3.
Time Frame: Up to 28 days
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants
  Alanine transaminase (ALT): Grade 0 | 3 | 0 | 3
  ALT: Grade 1 | 0 | 1 | 0
  Aspartate Aminotransferase (AST): Grade 0 | 3 | 1 | 3
  Bilirubin: Grade 0 | 3 | 1 | 3
  Creatinine: Grade 0 | 3 | 1 | 2
  Creatinine: Grade 2 | 0 | 0 | 1
  Hypoglycemia: Grade 0 | 3 | 1 | 3
  Hyperglycemia: Grade 0 | 3 | 1 | 3
  Hypokalemia: Grade 0 | 3 | 1 | 3
  Hyperkalemia: Grade 0 | 1 | 1 | 1
  Hyperkalemia: Grade 1 | 2 | 0 | 2
  Hyponatremia: Grade 0 | 3 | 1 | 3
  Hypernatremia: Grade 0 | 3 | 1 | 3
  Hemoglobin (Hb): Grade 0 | 2 | 1 | 2
  Hb: Grade 1 | 1 | 0 | 0
  Hb: Grade 2 | 0 | 0 | 1
  Absolute neutrophil count (ANC): Grade 0 | 2 | 1 | 0
  ANC: Grade 1 | 1 | 0 | 1
  ANC: Grade 3 | 0 | 0 | 1
  ANC: Grade 4 | 0 | 0 | 1
  Platelets: Grade 0 | 3 | 1 | 2
  Platelets: Grade 3 | 0 | 0 | 1

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of JNJ-63549109 (Metabolite of Lumicitabine)
Description: Cmax is the maximum observed plasma concentration of JNJ-63549109 (Metabolite of Lumicitabine).
Time Frame: Day 1 and Day 5
Population: Intent to Treat (ITT) set was defined as all randomized participants who receive at least 1 dose of study.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 1 | 3
nanogram/milliliter (ng/ml)
  Day 1 | 6184 | 7003 (3806)
  Day 5 | 3261 | 5112 (1665)

8. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) of JNJ-63549109 (Metabolite of Lumicitabine)
Description: AUC is the area under the plasma concentration-time curve of JNJ-63549109 (Metabolite of Lumicitabine).
Time Frame: Day 1 and Day 5
Population: ITT set was defined as all randomized participants who receive at least 1 dose of study.
Measure: Mean (Standard Deviation); unit: nanogram hour per milliliters (ng*h/ml)
Arm/Group | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 1 | 3
nanogram hour per milliliters (ng*h/ml)
  Day 1 | 12700 | 17800 (713.9)
  Day 5 | 11840 | 20500 (655.7)

9. Secondary Outcome: Trough Observed Analyte Concentration (C[Trough]) of JNJ-63549109 (Metabolite of Lumicitabine)
Description: C(trough) is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen of JNJ-63549109 (Metabolite of Lumicitabine).
Time Frame: Day 1 and Day 5
Population: ITT set was defined as all randomized participants who receive at least 1 dose of study.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 1 | 3
ng/ml
  Day 1 | 91.16 | 187.8 (52.97)
  Day 5 | 189.8 | 358.3 (37.42)

10. Secondary Outcome: Predicted Concentration of JNJ-63549109 (Metabolite of Lumicitabine) at 12 Hours Postdose (C12h)
Description: C12h is the predicted concentration of JNJ-63549109 at 12 hours Postdose. C12h is a model-based prediction. It was determined using a population pharmacokinetic (PK) model and based on the individual model predicted concentration-time profiles.
Time Frame: 12 hours postdose
Population: as for outcome 1
Arm/Group | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay is defined as the time from hospitalization to actual hospital discharge.
Time Frame: Up to 28 days
Population: Population included randomized or treated set. As the study was early terminated with fewer participants than planned, results for this endpoint could not be summarized. Hence, individual data for each participant was reported. Here, n (number analyzed) signifies specific participant evaluated in respective arm.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Hours
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 143.5 |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 | 167.8 |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 | 179.4 |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 |  | 167.8 |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1
  Participant 5 |  |  | 120
  Participant 6: number analyzed (Participants) | 0 | 0 | 1
  Participant 6 |  |  | 239.5
  Participant 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 7 |  |  | 149.3

12. Secondary Outcome: Number of Participants Admitted to the Intensive Care Unit (ICU)
Description: Number of participants who were admitted to the ICU was reported.
Time Frame: Up to 28 days
Population: Randomized or Treated set was defined as all participants who were in the Randomized Analysis Set (all randomized participants with a randomization date at or before the date of the first intake of medication, or with a randomization date and a missing date for first medication intake, analyzed as randomized) and/or the AST set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 0

13. Secondary Outcome: Duration of ICU Stay
Description: In the event that a participant required ICU, the duration for how long the participant remained in the ICU was reported.
Time Frame: Up to 28 days
Population: No participant was admitted to ICU hence results could not be determined for this outcome measure.
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Participants Who Required Supplemental Oxygen
Description: The number of participants who required supplemental oxygen above pre-RSV infection status was reported.
Time Frame: Up to 28 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 1 | 1 | 0

15. Secondary Outcome: Number of Participants Who Required Non-invasive Mechanical Ventilation Support
Description: The number of participants who required non-invasive mechanical ventilation support (that is, continuous positive airway pressure) above pre-RSV infection status was reported.
Time Frame: Up to 28 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Who Required Invasive Mechanical Ventilation Support
Description: The number of participants who required invasive mechanical ventilation support (for example, endotracheal-mechanical ventilation or mechanical ventilation via tracheostomy) above pre-RSV infection status was reported.
Time Frame: Up to 28 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 0

17. Secondary Outcome: Duration of Supplemental Oxygen
Description: Duration of supplemental oxygen above pre-RSV infection status was assessed.
Time Frame: Up to 28 days
Population: Population included randomized or treated set who received supplemental oxygen.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 1 | 1 | 0
Hours | 59.4 | 0.5 |

18. Secondary Outcome: Duration of Non-invasive Mechanical Ventilation Support
Description: Duration of non-invasive mechanical ventilation support (that is, continuous positive airway pressure) to deliver oxygen above pre-RSV infection status was measured.
Time Frame: Up to 28 days
Population: No participant received non-invasive mechanical ventilation support hence results could not be drawn for this outcome measure.
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Duration of Invasive Mechanical Ventilation Support
Description: Duration of invasive mechanical ventilation support (for example, endotracheal-mechanical ventilation or mechanical ventilation via tracheostomy) to deliver oxygen above pre-RSV infection status was measured.
Time Frame: Up to 28 days
Population: No participant received invasive mechanical ventilation support hence results could not be drawn for this outcome measure.
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Time to no Longer Requiring Supplemental Oxygen
Description: Time to no longer requiring supplemental oxygen above pre-RSV infection status was reported.
Time Frame: Up to 28 days
Population: Population included randomized or treated set who received supplemental oxygen.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 1 | 1 | 0
Hours | 59.4 | 0.5 |

21. Secondary Outcome: Time to Clinical Stability
Description: Time to clinical stability was defined as the time at which the following criteria are all met: normalization of blood oxygen level (return to baseline, by pulse oximetry) without the requirement of supplemental oxygen beyond baseline level, normalization of oral feeding, normalization of respiratory rate, and normalization of heart rate.
Time Frame: Up to 28 days
Population: Population included randomized or treated set. Due to early study termination and less number of participants collected data was not summarized. Hence, individual data for each participant was reported. Here, n (number analyzed) signifies specific participant evaluated in respective arm.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Hours
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 63.8 |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 | 39.5 |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 | 191.2 |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 |  | 63.3 |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1
  Participant 5 |  |  | 71.3
  Participant 6: number analyzed (Participants) | 0 | 0 | 1
  Participant 6 |  |  | 646.4
  Participant 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 7 |  |  | 0

22. Secondary Outcome: Time From Initiation of Study Treatment Until Peripheral Capillary Oxygen Saturation (SpO2) Greater Than or Equal to (>=)93 Percent (%) on Room Air Among Participants Who Were Not on Supplemental Oxygen Prior to Onset of Respiratory Symptoms
Description: Time from initiation of study treatment until SpO2 >=93% on room air among participants who were not on supplemental oxygen prior to the onset of respiratory symptoms was reported.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Time for Respiratory Rate to Return to Pre-RSV Infection Status
Description: Time for the respiratory rate to return to pre-RSV infection status was measured.
Time Frame: Up to 28 days
Population: Population included randomized or treated set. As study was terminated early with fewer participants than planned, results for this endpoint could not be summarized. Hence, individual data for each participant was reported. Here, n (number analyzed) signifies specific participant evaluated in respective arm.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Hours
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 0 |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 | 39.5 |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 | 46.4 |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 |  | 0 |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1
  Participant 5 |  |  | 71.3
  Participant 6: number analyzed (Participants) | 0 | 0 | 1
  Participant 6 |  |  | 646.4
  Participant 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 7 |  |  | 0

24. Secondary Outcome: Time for SpO2 to Return to Pre-RSV Infection Status
Description: Time for SpO2 to return to pre-RSV infection status was measured.
Time Frame: Up to 28 days
Population: Population included randomized or treated set. As study was terminated early with fewer participants than planned, data was not summarized. Hence, individual data for each participant was reported. Here, n (number analyzed) signifies specific participant evaluated in respective arm.
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Hours
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 0 |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 | 0 |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 | 70 |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 |  | 33.7 |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1
  Participant 5 |  |  | 0
  Participant 6: number analyzed (Participants) | 0 | 0 | 1
  Participant 6 |  |  | 0
  Participant 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 7 |  |  | 0

25. Secondary Outcome: Time for Body Temperature to Return To Pre-RSV Infection Status
Description: Time for body temperature to return to pre-RSV infection status was measured.
Time Frame: Up to 28 days
Population: as for outcome 24
Measure: Number; unit: Hours
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Hours
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 0 |  |
  Participant 2: number analyzed (Participants) | 1 | 0 | 0
  Participant 2 | 643.5 |  |
  Participant 3: number analyzed (Participants) | 1 | 0 | 0
  Participant 3 | 37.4 |  |
  Participant 4: number analyzed (Participants) | 0 | 1 | 0
  Participant 4 |  | 16.7 |
  Participant 5: number analyzed (Participants) | 0 | 0 | 1
  Participant 5 |  |  | 0
  Participant 6: number analyzed (Participants) | 0 | 0 | 1
  Participant 6 |  |  | 0
  Participant 7: number analyzed (Participants) | 0 | 0 | 1
  Participant 7 |  |  | 641.6

26. Secondary Outcome: Number of Participants With Acute Otitis Media
Description: Number of participants with acute otitis media was reported.
Time Frame: Up to 28 days
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 0

27. Secondary Outcome: Duration of Signs and Symptoms of RSV Infection
Description: Duration of signs and symptoms of RSV infection was assessed.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Severity of Signs and Symptoms of RSV Infection Assessed by the Pediatric RSV Electronic Severity and Outcome Rating System (PRESORS)
Description: The severity of signs and symptoms of RSV infection were assessed by the PRESORS. PRESORS Score consisted of 5-items, each score ranges from 0 to 3 and the total score was analyzed by summing up the individual score ranging from 0 (minimum; best) to 15 (maximum; worse).
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: RSV Viral Load Over Time
Description: RSV viral load over time was measured by qRT-PCR in the mid-turbinate nasal swab specimens.
Time Frame: On Day 2, 3, 4, 5, 6, 7, 10, 14 and 28
Population: Intention-To-Treat-infected (ITT-i) set was defined as all randomly assigned participants who receive at least 1 dose of study drug and who have an RSV infection confirmed by a polymerase chain reaction (PCR)-based assay at baseline or within 1 hour after the first study medication intake at the central laboratory.
Measure: Mean (Standard Deviation); unit: log10 per milliliters (log10/mL)
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
log10 per milliliters (log10/mL)
  Day 2 | 5.817 (2.2087) | 6.809 | 6.660 (0.9732)
  Day 3 | 5.443 (1.4645) | 6.000 | 5.351 (0.5794)
  Day 4 | 4.674 (2.4209) | 2.900 | 4.190 (1.4190)
  Day 5 | 3.808 (1.0049) | 5.949 | 4.521 (1.7506)
  Day 6 | 3.137 (1.9306) | 6.514 | 4.110 (1.6980)
  Day 7 | 2.994 (1.4450) | 4.584 | 2.754 (1.2688)
  Day 10 | 2.821 (1.5950) | 1.900 | 3.573 (0.7610)
  Day 14 | 1.900 (0.0000) | 2.900 | 1.983 (0.1443)
  Day 28 | 1.900 (0.0000) | 1.900 | 1.900 (0.0000)

30. Secondary Outcome: Peak Viral Load
Description: Peak viral load was measured by qRT-PCR in the mid-turbinate nasal swab specimens.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Time To Peak Viral Load
Description: Time to peak viral load was reported.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Percentage of Participants With Decline of Viral Load
Description: Percentage of participants with decline in viral load during treatment as measured by qRT-PCR was reported.
Time Frame: Up to 28 days
Population: ITT-i set was defined as all randomly assigned participants who receive at least 1 dose of study drug and who have an RSV infection confirmed by a PCR-based assay at baseline or within 1 hour after the first study medication intake at the central laboratory.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Percentage of participants | 100 | 100 | 100

33. Secondary Outcome: Time to RSV Ribonucleic Acid (RNA) Being Undetectable
Description: Time to RSV RNA being undetectable (the time from initiation of study treatment until the time at which it is observed that the virus is undetectable in an assessment and after which time no virus positive assessment follows) was assessed as measured by qRT-PCR.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

34. Secondary Outcome: Percentage of Participants With Undetectable RSV Viral Load
Description: Percentage of participants with the undetectable viral load was reported.
Time Frame: Up to 28 days
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: AUC of RSV RNA Viral Load From Baseline up to Day 10
Description: AUC of RSV RNA viral load was measured in mid-turbinate nasal swabs and in the endotracheal sample.
Time Frame: Baseline up to Day 10
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

36. Secondary Outcome: AUC of RSV RNA Viral Load From Baseline up to Day 14
Description: AUC of RSV RNA viral load was measured in midturbinate nasal swabs and in endotracheal samples.
Time Frame: Baseline up to Day 14
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: AUC of RSV Viral Load From Baseline Until 1 Day After the Last Dose of Study Drug
Description: AUC of RSV viral load was measured in midturbinate nasal swabs and in endotracheal samples.
Time Frame: Baseline Until 1 Day after the last dose of study drug (up to 10 days)
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With Emergent Postbaseline Changes in the RSV Polymerase L-gene and Other Regions of the RSV Genome Compared With Baseline Sequences
Description: Number of participants with emergent postbaseline changes in the RSV polymerase L-gene and other regions of the RSV genome compared with baseline sequences were reported.
Time Frame: Baseline up to 28 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 0

39. Secondary Outcome: Acceptability and Palatability of Lumicitabine Formulation as Assessed by Clinician Electronic Clinical Outcome Assessment (eCOA)
Description: Acceptability and Palatability of lumicitabine formulation was assessed by clinician eCOA questionnaire ranging from score 0 (minimum; best) to 8 (maximum; worse).
Time Frame: Up to Day 6
Population: as for outcome 1
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety analysis set included all participants who received at least 1 dose of drug.
Arm/Group | Placebo | Lumicitabine 40/20 mg/kg LD/MD | Lumicitabine 60/40 mg/kg LD/MD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Lumicitabine 40/20 mg/kg LD/MD (N=1) | Lumicitabine 60/40 mg/kg LD/MD (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Lumicitabine 40/20 mg/kg LD/MD (N=1) | Lumicitabine 60/40 mg/kg LD/MD (N=3)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Only 7 participants were treated before the study was prematurely terminated. Due to this small number of treated subjects, statistical analysis was not conducted as planned. Hence it was not possible to evaluate the primary or secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03333317/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT03333317/SAP_001.pdf